CLINICAL TRIAL: NCT00634790
Title: An Open-label Study to Assess the Safety and Tolerability of Xanax XR in the Treatment of Adolescents With Panic Disorder or Anxiety With Panic Attacks
Brief Title: A Study To Assess the Safety of Extended Release Alprazolam for the Treatment of Adolescents With Panic Disorder or Anxiety With Panic Attacks
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Please see Detailed Description for termination reason.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6131004
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder | interventions — Alprazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- alprazolam group (Active Comparator)
  Interventions: Drug: alprazolam XR

INTERVENTIONS:
Drug: alprazolam XR — Alprazolam XR oral tablet 1 mg daily for 7 days; thereafter the daily dose will be titrated at a maximum rate of 1 mg every 7 days up to a maximum dose of 6 mg; dose adjustments up or down may be made, at a rate not to exceed 1 mg every 7 days; alprazolam XR will be administered for a total of 6 months followed by a gradual taper at a rate of 1 mg every 7 days.
  Other Names: Xanax XR

SUMMARY:
The purpose of this study is to assess the long-term safety and tolerability of alprazolam extended release (XR) in adolescents with panic disorder, with or without agoraphobia, or in anxiety disorder with panic attacks. Efficacy, population pharmacokinetics of alprazolam XR and the relationship between alprazolam XR plasma concentrations and efficacy outcomes will also be evaluated.

DETAILED DESCRIPTION:
Due to recruitment difficulties in this adolescent population, the clinical program for alprazolam XR was cancelled and this study was terminated on 1 September 2004. There were no safety concerns that led to this decision.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet one of the following 6 diagnoses: a. A current diagnosis of panic disorder with or without agoraphobia; b. Generalized anxiety disorder with a history of at least one panic attack in the course of their illness; c. Social anxiety disorder (social phobia) with a history of at least one panic attack in the course of their illness; d. Separation anxiety with a history of at least one panic attack in the course of their illness; e. Posttraumatic stress disorder with a history of at least one panic attack in the course of their illness; f. Anxiety not otherwise specified with a history of at least one panic attack in the course of their illness.
* Educational level, intelligence, or other mental condition in the subject and/or his/her parent(s) are judged by the investigator to be sufficient to permit adequate informed consent/assent to be obtained, and for study procedures to be complied with.

Exclusion Criteria:

* Current (in the past 6 months) diagnosis of obsessive compulsive disorder, major depressive disorder, dysthymic disorder, or alcohol and/or substance dependence.
* Current (in the past 3 months) diagnosis of alcohol and/or substance abuse.
* Primary diagnosis of conduct disorder, oppositional defiant disorder, or Attention Deficit Hyperactivity Disorder.
* Any current or past history of schizophrenia or psychosis; bipolar disorder or cyclothymia; dementia, delirium or other organic brain disease; an eating disorder; mental retardation, Asperger's disorder, or any other serious developmental disorder.
* A Childhood Depression Rating Scale, Revised score >35.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2004-05; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Endpoint change from baseline to Week 24 in Digit Symbol-Coding Test, immediate recall, and delayed recall | 24 weeks
Baseline-to-peak Physician's Withdrawal Checklist change score during 6-week taper off alprazolam | 6 week taper
The incidence of treatment-emergent adverse event during treatment with alprazolam XR | 24 weeks with taper

SECONDARY OUTCOMES:
Descriptive estimates of the persistence of safety events and adverse events at study endpoint | 24 weeks with taper
Endpoint change from baseline to Week 24 in the Panic Disorder Severity Scale-Adolescent version total and item scores | 24 weeks
Endpoint (Week 24) Clinical Global Impression (CGI)-Improvement score | 24 weeks
Endpoint change from baseline to Week 24 in CGI-Severity score | 24 weeks
Endpoint (Week 24) Pediatric Quality of Life, Enjoyment, and Satisfaction Questionnaire improvement score | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (46):
- United States (46):
  - Pfizer Investigational Site, Little Rock, Alaska
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Burbank, California
  - Pfizer Investigational Site, El Centro, California
  - Pfizer Investigational Site, La Mesa, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Oceanside, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Marcos, California
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Hialeah, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, North Miami, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Schaumburg, Illinois
  - Pfizer Investigational Site, Terre Haute, Indiana
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Owensboro, Kentucky
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Clinton Township, Michigan
  - Pfizer Investigational Site, Saint Paul, Minnesota
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Clementon, New Jersey
  - Pfizer Investigational Site, Kenilworth, New Jersey
  - Pfizer Investigational Site, Morristown, New Jersey
  - Pfizer Investigational Site, Bismarck, North Dakota
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Lyndhurst, Ohio
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Bala-Cynwyd, Pennsylvania
  - Pfizer Investigational Site, Hershey, Pennsylvania
  - Pfizer Investigational Site, Media, Pennsylvania
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Selmer, Tennessee
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Midlothian, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Middleton, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6131004&StudyName=A%20Study%20To%20Assess%20the%20Safety%20of%20Extended%20Release%20Alprazolam%20for%20the%20Treatment%20of%20Adolescents%20with%20Panic%20Disorder%20or%20Anxiety%20with%20Pan